CLINICAL TRIAL: NCT00452842
Title: An Observational Safety Follow Up Trial Of The Occurrence Of Major Cardiovascular Events And All Cause Mortality In Subjects Who Participated In Selected Torcetrapib/Atorvastatin Clinical Trials.
Brief Title: Safety FollowUp Study Of Cardiovascular Events In Subjects Who Participated In Selected Torcetrapib/Atorvastatin Studies
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Other Study IDs: A5091075
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2007-12

CONDITIONS: Cardiovascular Disease; Cerebrovascular Disorders
MeSH Terms: conditions — Cardiovascular Diseases; Cerebrovascular Disorders

SUMMARY:
An observational safety follow up trial will be conducted to monitor the occurrence of cardiovascular events and all cause mortality in subjects who participated in selected torcetrapib/atorvastatin Phase 1, 2, and 3 clinical trials. No hypotheses will be tested.

DETAILED DESCRIPTION:
Study A5091075, an observational study in subjects who had previously been treated with torcetrapib, was terminated on 20 Dec 2007. The study was terminated following reviews of final safety information from prior torcetrapib studies and the low participation rates observed during the recruitment period for study A5091075 . On the basis of this new information the Sponsor determined that it was unlikely that this study would result in new and scientifically valid information.

ELIGIBILITY:
Inclusion Criteria:

* Have signed informed consent prior to the initiation of any study-specific activities.
* Have participated in selected torcetrapib/atorvastatin Phase 1, 2, and 3 clinical trials and were treated with randomized study medication.

Exclusion Criteria:

* There are no exclusion criteria.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26784
Dates: Start 2007-10

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Clearwater, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5091075&StudyName=Safety%20FollowUp%20Study%20Of%20Cardiovascular%20Events%20In%20Subjects%20Who%20Participated%20In%20Selected%20Torcetrapib/Atorvastatin%20Studies